CLINICAL TRIAL: NCT06518512
Title: Automated Vision Assessment and Impairment Detection Through Gaze Analysis in Wet Age Related Macular Degeneration (AMD) Patients: a Prospective Clinical Evaluation (AVIGA2)
Brief Title: Automated Vision Assessment and Impairment Detection Through Gaze Analysis in Wet AMD Patients
Acronym: AVIGA2
Status: Active, not recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Occutrack Medical Solutions Pte Ltd (Unknown)
Responsible Party: Principal Investigator, Laude Augustinus, Adj A/Prof Laude Augustinus, Tan Tock Seng Hospital
Other Study IDs: 2022/00600
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration; Wet Age-related Macular Degeneration
Keywords: AMD; wet AMD; wAMD; PCV; macular degeneration; gaze analysis
MeSH Terms: conditions — Macular Degeneration | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AVIGA2: Eye gaze tracking using the AVIGA tool
  Interventions: Device: Automated Vision Assessment and Impairment Detection through Gaze Analysis (AVIGA) system

INTERVENTIONS:
Device: Automated Vision Assessment and Impairment Detection through Gaze Analysis (AVIGA) system — AVIGA is an automated method and system for vision assessment of a subject. The method includes the following: determining a set of test patterns for the subject based on a preliminary assessment of an eye of the subject; displaying the set of test patterns sequentially to the subject; collecting data on the subject's gaze in response to each test pattern displayed; and correlating central vision function of the subjects to the collected gaze data.
  Subjects perform the AVIGA test monocularly and pursue a pre-determined target moving in a customized waveform across the computer screen. The trail of the gaze points generated by the subject following the target is simultaneously recorded and stored.
  1. Static Fixation Evaluation (SFE)
  2. Static Perimetry Assessment (SPA)
  3. Static Perimetry Sensitivity Assessment (SPSA)
  4. Pursuit

SUMMARY:
The study aims to evaluate the Automated Vision Assessment and Impairment Detection through Gaze Analysis (AVIGA) system in the ability to detect and assess central vision dysfunction in a personalized, adaptive, objective, and automated way through eye gaze tracking in age-related macular degeneration (AMD). We also aim to develop a novel algorithm / scoring methodology for disease activity monitoring over time (delta-change). AVIGA visual risk prediction cut-off scores will be presented together with probabilities of occurrence of prespecified adverse clinical outcome.

DETAILED DESCRIPTION:
Macula degeneration is more prevalent with ageing and can result in blurred or distorted vision, often accompanied by a dark patch blocking the center of the visual field. In the management of age-related macular degeneration (AMD), patients are required to attend regular check-ups at the specialist eye clinic by the clinician to monitor if their disease. The eye examinations that patients undergo during these clinic visits which may include fundoscopy and optical coherence tomography. A preventive treatment for exudative or wet AMD is the administration of an intravitreal injection of an anti-vascular endothelial growth factor (anti- VEGF) at these regular clinic sessions. Although anti-vascular endothelial growth factor (VEGF) injections are an effective treatment for many patients with Wet-AMD, there are several unmet needs in treatment of AMD and none of them cures the disease or reverses its course. Some patients do not respond to VEGF injections. There are no standardized treatment schedules, there is a large treatment burden, and visual loss continues over time. Additionally, the main drawback of anti-VEGF therapy is its high cost, which suppose a significant burden on health systems, and often makes such a regimen unaffordable in clinical practice.

There is no treatment for GA. Therefore, the prevention of advanced disease like Wet-AMD and finding new and effective treatments remain a significant challenge. Advances in imaging and genetics and molecular technologies have led to the identification of new risk factors for disease progression, but not all have been evaluated in comprehensive prediction models. Perhaps, comprehensive prediction models could lead to the development of tailored, individualized therapy and improve the personalised healthcare.As such, the application of this Novel OCCUTRACK Technology to develop a comprehensive risk score algorithm and to estimate the risk scores to identify individuals at high risk for disease progression to advanced stages would result in earlier intervention and reduced burden of visual loss due to AMD. This approach could enable the tailored individualized Anti-VEGF Therapy to promote personalized medicine and improve the quality of life of patients with Wet-AMD. A Proof-of-Concept (POC) was completed by TTSH clinician and AStar-I2R scientist to co-develop and patent a software - Automated Vision Assessment and Impairment Detection through Gaze Analysis (AVIGA). A local medical incubator, Trendlines Medical Singapore, has licensed it from the research party. This led to the spin-off of a new company - Occutrack Pte Ltd to continue the collaboration with TTSH, focusing on the commercialization of the AVIGA. The AVIGA system incorporates an ocular tracking system with gaze tracking algorithms designed to provide a comprehensive assessment of a patient's vision. With this non-invasive technology, retinal specialists can monitor the real time progression and prognosis of patients with AMD while they are in the comfort of their own home without the need for manual or skilled intervention and expensive equipment. This project proposal is to evaluate the performance and accuracy of the AVIGA technology as a tool for determining AMD disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the age group = 55 years and above.
* Both genders
* Subjects with Wet-AMD
* Ability to comply with the study protocol, in the investigator's judgment
* Subjects must be able to understand and provide informed consent. A signed informed consent form must be provided before any study assessments are done.

Exclusion Criteria:

* Uncontrolled blood pressure, defined as systolic blood pressure >180 millimeters of mercury (mmHg) and/or diastolic blood pressure >100 mmHg while a patient is at rest.
* Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid in the study eye
* Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active ocular inflammation or suspected or active ocular or periocular infection in either eye
* Other protocol-specified exclusion criteria may apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders aged 55 years and above diagnosed with wet AMD. Participants recruited must be cognitively coherent.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between AVIGA and standard clincial measures for detecting AMD activity | 1 year
  Assessment of the agreement between AVIGA-derived eye gaze tracking metrics and standard clinical measures of central visual function (optical coherence tomography [OCT], visual acuity, and fundoscopy) in detecting active aged-related macular degeneration (AMD). This outcome will determine whether AVIGA can serve as a reliable tool to detect AMD disease repeatability.

SECONDARY OUTCOMES:
Development and validation of an AVIGA Algorithm for tracking AMD progression | 1 year
  Evaluation of a new AVIGA algorithm to detect longitudinal changes in visual function and disease activity in AMD patients. The algorithm's outputs will be compared against changes observed in OCT, visual acuity, and fundus imaging over time. This outcome will assess the algorithm's ability to track disease progression and treatment response quantitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Augustinus Laude, MBChB, Principal Investigator — Tan Tock Seng Hospital; Zheng Kuang Noel Soh, BSc, Study Director — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huiying Liu, Wong D, Ai Ping Yow, Yanwu Xu, Fengshou Yin, Laude A, Tock Han Lim. Determining the difference in eyegaze measurements in individuals with age related macular degeneration. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:1348-1351. doi: 10.1109/EMBC.2016.7590957. PMID 28268575
- [Result] Huiying Liu, Yanwu Xu, Damon Wong, Ai Ping Yow, Laude A, Tock Han Lim. Detecting impaired vision caused by AMD from gaze data. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:3142-3145. doi: 10.1109/EMBC.2017.8037523. PMID 29060564
- [Result] Age-Related Eye Disease Study Research Group. The Age-Related Eye Disease Study (AREDS): design implications. AREDS report no. 1. Control Clin Trials. 1999 Dec;20(6):573-600. doi: 10.1016/s0197-2456(99)00031-8. PMID 10588299
- [Result] Chew EY, Clemons TE, Agron E, Sperduto RD, Sangiovanni JP, Davis MD, Ferris FL 3rd; Age-Related Eye Disease Study Research Group. Ten-year follow-up of age-related macular degeneration in the age-related eye disease study: AREDS report no. 36. JAMA Ophthalmol. 2014 Mar;132(3):272-7. doi: 10.1001/jamaophthalmol.2013.6636. PMID 24385141
- [Result] AREDS2 Research Group; Chew EY, Clemons T, SanGiovanni JP, Danis R, Domalpally A, McBee W, Sperduto R, Ferris FL. The Age-Related Eye Disease Study 2 (AREDS2): study design and baseline characteristics (AREDS2 report number 1). Ophthalmology. 2012 Nov;119(11):2282-9. doi: 10.1016/j.ophtha.2012.05.027. Epub 2012 Jul 26. PMID 22840421
- [Result] AREDS2-HOME Study Research Group; Chew EY, Clemons TE, Bressler SB, Elman MJ, Danis RP, Domalpally A, Heier JS, Kim JE, Garfinkel R. Randomized trial of a home monitoring system for early detection of choroidal neovascularization home monitoring of the Eye (HOME) study. Ophthalmology. 2014 Feb;121(2):535-44. doi: 10.1016/j.ophtha.2013.10.027. Epub 2013 Nov 8. PMID 24211172
- [Result] Mathew R, Sivaprasad S. Environmental Amsler test as a monitoring tool for retreatment with ranibizumab for neovascular age-related macular degeneration. Eye (Lond). 2012 Mar;26(3):389-93. doi: 10.1038/eye.2011.326. Epub 2011 Dec 16. PMID 22173073
- [Result] Ai Ping Yow, Damon Wong, Huiying Liu, Hongyuan Zhu, Ivy Jing-Wen Ong, Laude A, Tock Han Lim. Automatic visual impairment detection system for age-related eye diseases through gaze analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:2450-2453. doi: 10.1109/EMBC.2017.8037352. PMID 29060394
- [Result] Trevino R, Kynn MG. Macular function surveillance revisited. Optometry. 2008 Jul;79(7):397-403. doi: 10.1016/j.optm.2007.09.017. PMID 18577497
- [Result] Kawasaki R, Wang JJ, Aung T, Tan DT, Mitchell P, Sandar M, Saw SM, Wong TY; Singapore Malay Eye Study Group. Prevalence of age-related macular degeneration in a Malay population: the Singapore Malay Eye Study. Ophthalmology. 2008 Oct;115(10):1735-41. doi: 10.1016/j.ophtha.2008.02.012. Epub 2008 Apr 25. PMID 18439679
- See also: Vision assessment based on gaze US20190110678A1 — https://patents.google.com/patent/US20190110678A1/en
- See also: The significance of early detection of age-related macular degeneration: Richard & Hinda Rosenthal Foundation lecture, The Macula Society 29th annual meeting. — https://europepmc.org/article/MED/17891011